CLINICAL TRIAL: NCT02436525
Title: Faculty of Dental Medicine, Boys, Cairo Al-Azhar University
Brief Title: Microbial and Periodontal Changes Associated With Conventional Versus Self Ligating Brackets
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Esam Al-hendi, Head of Dental department in Jepleh Hospital, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 005OR.
Record Dates: First submitted 2015-04-19; First posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-02

CONDITIONS: Pocket Depth; Plaque Accumulation; Gigival Bleeding

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group I: (Active Comparator): will be treated using conventional stainless steel orthodontic brackets ligated with stainless steel ligature. Oromco - USA.
  .
  Interventions: Device: conventional stainless steel orthodontic brackets ligated with stainless steel ligature (Oromco - USA)
- Group II (Experimental): : will be treated using passive self-ligating stainless steel orthodontic brackets Oromco - USA.
  Interventions: Device: passive self-ligating stainless steel orthodontic brackets (Oromco - USA)
- Group III: (Experimental): will be treated by active self-ligating stainless steel orthodontic brackets Oromco - USA .
  Interventions: Device: active self-ligating stainless steel orthodontic brackets (Oromco - USA)

INTERVENTIONS:
Device: conventional stainless steel orthodontic brackets ligated with stainless steel ligature (Oromco - USA)
  Other Names: conb
  Arms: Group I:
Device: passive self-ligating stainless steel orthodontic brackets (Oromco - USA)
  Other Names: pasb
  Arms: Group II
Device: active self-ligating stainless steel orthodontic brackets (Oromco - USA)
  Other Names: actb
  Arms: Group III:

SUMMARY:
Microbial and periodontal changes associated with conventional versus self ligating brackets.

The aim of this study will be to compare microbial and periodontal changes associated with conventional versus self ligating brackets.

DETAILED DESCRIPTION:
Microbial and periodontal changes associated with conventional versus self ligating brackets.

Protocol submitted in partial fulfillment for the requirements of Master Degree in Orthodontics

Accumulation of biofilm on the tooth surfaces is associated with increased levels of oral streptococcus mutans and lactobacilli, which have been proved to be responsible for the onset of enamel demineralization and periodontal disease.

It has been shown that fixed appliance provides large number of retentive areas for plaque accumulation and impedes oral hygiene.

Three methods are currently used to connect the arch wire to the brackets, which are : ligation with stainless steel ligatures , using elastomeric ligatures, and the self-ligating brackets. , Each of these method has it's advantages and disadvantages, concerning the biofilm retention and the level of microorganisms. , Orthodontic treatment with conventional brackets my presents some periodontal changes caused by difficulty in oral hygiene maintenance, greater accumulation and qualitative alteration of plaque. Thus, in order to control oral hygiene and plaque level during fixed appliance therapy, manufacturers introduced self-ligating brackets (SLBs) which have been claimed to provide better oral hygiene and less plaque accumulation, because of fewer retentive sites for microbial colonization; without the need for stainless steel and elastomeric ligature. Clinically, the side effects of fixed orthodontic treatment, such as the qualitative bacterial shift, are manifested as plaque associated gingivitis, an increase in pocket probing depth (PPD), and bleeding on probing.

Fewer studies have compared conventional and self-ligating brackets in relation to oral hygiene, microbial count and periodontal indices. Therefore, the present study will be conducted to evaluate and compare microbial and periodontal changes with conventional and self ligating brackets.

The aim of this study will be to compare microbial and periodontal changes associated with conventional versus self ligating brackets.

Subjects and method

Study design:

Randomized controlled clinical trial

Study setting and population:

The sample of this study will be consisted of forty five patients selected from Outpatient Clinic, Orthodontic Department, Faculty of Dental Medicine, Boys, Cairo, Al-Azhar University.

Interventions:

The patients will be divided randomly into three groups and will be treated separately as follows:

* Group I: will be treated using conventional stainless steel orthodontic brackets ligated with stainless steel ligature.
* Group II: will be treated using passive self-ligating stainless steel orthodontic brackets.
* Group III: will be treated by active self-ligating stainless steel orthodontic brackets.

Records:

For all patients the following records will be taken before and after treatment:

1. Standardized Orthodontic study cast.
2. Standardized intra oral and extra oral photographs.
3. Standardized panoramic radiograph.
4. Standardized lateral cephalometric radiograph.

Observations:

• Periodontal parameters: The following clinical parameters will be recorded at baseline before treatment and at monthly interval for 6 months after bonding;

1. Pocket probing depth .
2. Plaque index (Silness and Loe) .
3. The presence or absence of bleeding on probing .

   * Microbial parameters:

Plaque sample will be taken at base line and at monthly interval for six months after bonding. The sample will be taken from the maxillary left canine, second premolar and the right central incisor and the mandibular right canine, second premolar and the left central incisor.

Plaque sample will be send to laboratory for isolation of streptococcus mutans and lactobacilli. The isolated strains will be cultured and counted.

Ethical consideration:

All patients will clearly understand the purpose of the study and give their consent by signing an informed consent (attached copy of the consent form).

Patient's instructions:

Instructions form (a copy attached) will be signed by all patients and their parents before commencing the study.

Data management and analysis:BN All the obtained results will be gathered and statistically analyzed using Statistical Package for Social Sciences (SPSS, version 16, Inc., Chicago, Ill).

ELIGIBILITY:
Inclusion Criteria:

All patients should satisfy the following criteria:

1. Age ranged between 14-18 years.
2. All permanent teeth erupted (excluding third molars).
3. Angle Class I with normal facial proportion.
4. Moderate crowding (from 4 to 6 mm) or irregularity index greater than 4.
5. All cases require treatment with fixed appliance with non extraction approach.
6. Good oral and general health.
7. No previous or current periodontal diseases.
8. No systemic disease or medication that may interfere with orthodontic teeth movement.
9. No history of trauma, bruxism or parafunction.
10. No previous orthodontic treatment.

Exclusion Criteria:

1. Abnormal anteroposterior relationship or steep mandibular plane.
2. Crowding more than 6 mm.
3. Poor oral hygiene or periodontal affection.
4. Uncooperative patients.
5. Smoker patients.
6. Pregnant females.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Pocket depth | every month for six months
  Pocket depth measured by a Williams periodontal probe at baseline before treatment and at monthly interval for 6 months after bonding.
plaque accumulation | every month for 6 months after bonding.
  plaque accumulation will be assess using Silness and Loe index
Gingival bleeding | every month for 6 months after bonding.
  Gingival bleeding will be evaluated by the presence or absence of bleeding on probing
Composite measure of Microbial parameters | every month for 6 months after bonding.
  Plaque sample will be taken at base line and at monthly interval for six months after bonding Plaque sample will be send to laboratory for isolation of streptococcus mutans and lactobacilli. The isolated strains will be cultured and counted

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Cairo Governorate, Egypt